CLINICAL TRIAL: NCT01236898
Title: Pharmacokinetic Study on N-acetylneuraminic Acid in Patients With Distal Myopathy With Rimmed Vacuoles (DMRV) - Hereditary Inclusion Body Myopathy (hIBM)
Brief Title: Pharmacokinetic Study on N-acetylneuraminic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tohoku University (Other)
Responsible Party: Tohoku University Hospital Internal Neurology, Tohoku University Hospital Internal Neurology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sialic acid-1
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-08

CONDITIONS: Nonaka Myopathy; Hereditary Inclusion Body Myopathy
Keywords: N-acetylneuraminic acid,; pharmacokinetics; hIBM
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NPC-09 (Experimental): Period 1: NPC-09 800mg single oral dosing NPC-09 800mg three times oral dosing a day Period 2: NPC-09 800mg three times oral dosing a day for 5 consecutive days
  Interventions: Drug: NPC-09

INTERVENTIONS:
Drug: NPC-09 — NPC-09 tablet NPC-09 contains 50mg or 100mg N-acetylneuraminic acid (anhydride)

SUMMARY:
The aim of this study is to investigate pharmacokinetics and safety of N-acetylneuraminic acid in patients with Distal myopathy with rimmed vacuoles (DMRV) - hereditary inclusion body myopathy (hIBM). Dosages are 800mg single and three times a day and 800mg 3 times a day for 5 consecutive days. N-acetylneuraminic acid and N-glycolylneuraminic acid in serum and urine are measured before and after oral administration of N-acetylneuraminic acid.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed mutations in GNE gene
* No severe complications when informed consent is obtained
* More than 40 kg in weight before administration

Exclusion Criteria:

* Hepatic laboratory parameters (AST, ALT, γ-GTP) or Renal laboratory parameters (Cr, BUN) are greater than three times of upper limit of reference value
* Presence or history of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, gastrointestinal, brain, psychiatric, neurologic disease
* Intake of supplement contains sialic acid, St. John's wort or grapefruit within 7 days
* Enrollment in another investigational study within 3 months
* More than 400 mL blood donation within 3 months
* Presence of alcohol or drug dependency
* Women who are pregnant , breast feeding or possible to be pregnant.
* Patients whom the investigator judges not to be appropriate for the subject

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in serum concentration of N-acetylneuraminic acid | 24 hours before dosing and dosing days
  Patients with DMRV(hIBM) show low serum N-acetylneuraminic acid level.
Change in pharmacokinetic parameters of N-acetylneuraminic acid: AUCt | 24 hours before dosing and dosing days
Change in amount of urinary excretion of N-acetylneuraminic acid | 24 hours before dosing and dosing days
Safety(adverse events) | Up to 5-7 days after dosing

SECONDARY OUTCOMES:
Change in serum concentration of N-glycolylneuraminic acid | 24 hours before dosing and dosing days
Change in pharmacokinetic parameters of N-glycolylneuraminic acid: AUCt | 24 hours before dosing and dosing days
Change in amount of urinary excretion of N-glycolylneuraminic acid | 24 hours before dosing and dosing days

CONTACTS AND LOCATIONS:
Overall Officials: Masashi Aoki, Principal Investigator — Tohoku University Hospital Internal Neurology
Locations (1):
- Tohoku University Hospital, Sendai, Miyagi, Japan